CLINICAL TRIAL: NCT04626843
Title: Feasibility Study of Intermittent Fasting in Chronic Lymphocytic Leukemia and Small Lymphocytic Lymphoma (CLL/SLL) Patients at BC Cancer- Victoria
Brief Title: Intermittent Fasting and CLL/SLL
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Eleah Stringer (Other)
Collaborators: BC Cancer Foundation (Other)
Responsible Party: Sponsor-Investigator, Eleah Stringer, Oncology Dietitian, British Columbia Cancer Agency
Organization: British Columbia Cancer Agency (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H19-03702
Record Dates: First submitted 2020-09-30; First posted 2020-11-13 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-02

CONDITIONS: Neoplasms; Leukemia, Lymphocytic, Chronic; Lymphoma, Small Lymphocytic; Intermittent Fasting; Diet Habit; Inflammation
MeSH Terms: conditions — Neoplasms; Leukemia, Lymphocytic, Chronic, B-Cell; Intermittent Fasting; Feeding Behavior; Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intermittent fasting (Experimental)
  Interventions: Other: Intermittent fast

INTERVENTIONS:
Other: Intermittent fast — 16/8 fasting method: fast for 16 hours of the day with an 8 hours feeding window for a duration of 3 months.

SUMMARY:
What are the investigators trying to do? By most measures, humans consume more food than needed. Over several decades, overconsumption has led to an increase in a number of diseases, including cancer. What if this could be reversed, or slowed down, by fasting? Would that improve how cancer patients respond to chemotherapy? Could simply changing eating patterns to reduce overall intake be a way to prevent and/or manage cancer? All of these are important questions and the investigators are undertaking a new initiative to study how nutrition and dietary behaviours affect cancer patients.

Fasting: A way to improve overall health and increase our defenses to cancer Fasting in various forms has been shown to have a number of health benefits. Intermittent fasting, or time restricted feeding, has been shown to reverse or improve various diseases such as diabetes, heart disease and metabolic syndrome, decrease the risk of cancer, and significantly extend the life of an individual. In previous studies, fasting was well-tolerated with notable improvements in energy levels, sense of well-being, and sleep quality. In cancer patients, clinical trials have demonstrated intermittent fasting to lessen some of the short-term side effects of chemotherapy such as nausea, fatigue, and sleep quality. How fasting alters the course of cancer or improve immune defenses is not yet known but may be an alternative way to treat or manage cancer.

The study plan The investigators plan to examine the effects of intermittent fasting (time restricted feeding) in patients with chronic lymphocytic leukemia (CLL). CLL is the most common chronic leukemia and is presently incurable. The advantage of choosing this patient population is that the cancer is easily assessed with a blood test measuring the amount of cancerous white cells (lymphocytes). Patients who consent to participate in this study will, through the support of an oncology dietitian and after a period of transition, split their daily feeding into a fasting period and a non-fasting period. This regime is as simple as skipping or having a late breakfast. At this time, participants will not be required to limit their total caloric intake.

What is required from the participant? The investigators will assess whether intermittent fasting reduces the cancer by measuring the lymphocyte count in the blood over a period of 3 months. Study participants will complete questionnaires to help determine if fasting causes any change in their quality of life. The effects of intermittent fasting on a cancer control system called autophagy, as well as its effects on inflammation will be studied in the Deeley Research Centre laboratory at BC Cancer.

What is the short- and long-term impact? In the short-term, if intermittent fasting can have an effect cancer lymphocyte count or on autophagy, then investigators will proceed with further studies to try and optimize the effects of intermittent fasting. In the long-term, this study is expected to be the first-ever to shed light on how intermittent fasting may be linked to cancer survival and/or growth. If true, this will open up new avenues to re-evaluate the inclusion of diet into cancer treatment protocols.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of CLL or SLL
* Age </=85
* Lymphocytes >/=40 and <150
* Hemoglobin >/=100g/L
* Platelet >100 x 10*9/L
* BMI of >/= 20kg/m2
* Eastern Cooperative Oncology Group (ECOG) Performance Status </=2
* Not on anti-lymphoma therapy within the past 3 months
* Not receiving anti-lymphoma therapy and not expected to require initiation of anti-lymphoma therapy within the next 3 months

Exclusion Criteria:

* Patient unable to give consent
* Patient on medications required to be taken with food during the fasting window
* Pregnancy
* Diabetes mellitus
* BMI drop to </= 18.5kg/m2 at any time during study

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2021-02-03 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in lymphocyte count | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in lymphocyte count will be measured between each peripheral blood draw.
Change in quality of life | Pre-intervention, day 90 of intervention, 1 month post-intervention
  A quality of life questionnaire, European Organization for Research and Treatment of Cancer Quality of Life Questionnaire Cancer 30 (EORTC QLQ-C30) version 3, will be administered to assess to subjective changes in well-being. It comprises 30 items (i.e. single questions), 24 of which are aggregated into nine multi-item scales, that is, five functioning scales (physical, role, cognitive, emotional and social), three symptom scales (fatigue, pain and nausea/vomiting) and one global health status scale. The remaining six single-item scales assess symptoms. All of the scales and single-item measures range in score from 0 to 100. Higher score for the functioning scales and global health status denote a better level of functioning (i.e. a better state of the patient), while higher scores on the symptom and single-item scales indicate a higher level of symptoms (i.e. a worse state of the patient).
Change in inflammation | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in c-reactive protein (CRP) will be measured between each peripheral blood draw.
Change in metabolic profiles | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Changes in metabolomic profiles will be measured between each peripheral blood draw.
Change in autophagy status | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  This includes standard flow cytometric analysis of lymphocyte subsets: a panel established by the Human Immunology Consortium Project as well as additional in-house markers to enumerate the frequency of lymphocytes before and at various time points post-treatment. The extent of autophagy will be tested by performing cytometry and western blotting assays using LC3II and p62 as readouts. Total cell counts in different lymphocyte subsets including, but not limited to, cluster of differentiation (CD) 3, CD8, CD4, CD20, CD19, and forkhead box P3 (FoxP3) will be assayed in conjugation with glucose uptake and mitochondrial function.
Immune cell gene expression profiles | Within 3 months pre-intervention, monthly during intervention, 1 month post-intervention
  Expression profiles of selected immune cell genes

SECONDARY OUTCOMES:
Change in gut microbiome (optional) | 1 month pre-intervention, day 30 of intervention, day 90 of intervention
  Stool samples to identify baseline and fasting-induced changes in abundance and repertoire of the gut microbiota

CONTACTS AND LOCATIONS:
Locations (1):
- Eleah Stringer, Victoria, British Columbia, Canada

IPD SHARING:
Plan to Share IPD: No